CLINICAL TRIAL: NCT04028349
Title: An Open-label, Single Arm Study to Provide Additional Information on Immunogenicity and Safety of Ad26.ZEBOV/MVA-BN-Filo
Brief Title: ZEBOVAC (Ebola Vaccine Trial, Ad26.ZEBOV/MVA-BN-Filo)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Collaborators: Epicentre, Mbarara, Uganda (Unknown); Janssen Pharmaceutica N.V., Belgium (Industry); Coalition for Epidemic Preparedness Innovations (Other); Epicentre, Paris, France. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RGPK181201
Record Dates: First submitted 2019-07-03; First posted 2019-07-22 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Ad26.ZEBOV/ MVA-BN-Filo Vaccines
  Interventions: Drug: Ad26.ZEBOV/MVA-BN-Filo

INTERVENTIONS:
Drug: Ad26.ZEBOV/MVA-BN-Filo — Candidate Ebola Vaccine

SUMMARY:
An open-label, single arm phase II study of the candidate Ebola Vaccine Ad26.ZEBOV/MVA-BN®-Filo

DETAILED DESCRIPTION:
This is an interventional, single arm, open-label, non-randomized, phase II study to accumulate additional data on immunogenicity and safety of Ad26.ZEBOV/MVA-BN®-Filo against Ebola virus disease.

It also has a qualitative component to better understand knowledge about Ebola virus disease and the perception and attitudes towards the vaccine amongst participants (Healthcare and Frontline workers).

ELIGIBILITY:
Inclusion criteria Each potential participant must satisfy all of the following criteria to be enrolled in the study.

1. Each participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study. In case the participant cannot read or write, the procedures must be explained and informed consent must be witnessed by a literate third party not involved with the conduct of the study.
2. Participant must be a man or woman aged 18 years or older, inclusive at day of signing the ICF.
3. Healthcare or frontline workers within Mbarara district:

   * Healthcare workers such as physicians, clinicians, nurses, nurse aides, laboratory personnel, pharmacists, village health teams etc...
   * Frontline workers such as cleaners, mortuary attendants, security staff, receptionists and outside structure's staff deployed in the response (surveillance team, ambulance team, burial or worker responsible for swabbing deceased persons)
   * Healthcare staff and medical students or other students undertaking a health related course providing non-Ebola related care which places them in contact with patients at public and private health centres or clinics
4. Participant must be healthy in the investigator's clinical judgment on the basis of medical history, physical examination and vital signs performed at screening. If any of the assessed parameters (such as vital sign or laboratory value) is abnormal (and considered clinically significant by the investigator), it may be re-assessed only once at a later time point within the screening window (7 days) to determine eligibility.
5. Before enrolment (on Day 1), a sexually active woman must be either:

   Of childbearing potential and practicing a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for participants participating in clinical studies, beginning at least 28 days prior to vaccination.

   OR Not of childbearing potential: postmenopausal (>45 years of age with amenorrhea for at least 2 years); permanently sterilized (eg, bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy); or otherwise be incapable of pregnancy.

   Note: If the social situation of a woman changes after start of the study (eg, woman who is not heterosexually active becomes active), she must begin a highly effective method of birth control, as described above.
6. A woman of childbearing potential must have a negative urine β-human chorionic gonadotropin (β-hCG) pregnancy test at screening and a negative urine β-hCG pregnancy test immediately prior to each study vaccine administration.

   Note: If the pregnancy test result is positive, in order to maintain participant confidentiality, the investigator will ensure adequate counseling and follow-up will be made available.
7. Participant must be available and willing to participate for the duration of the study visits and follow-up.
8. Participant must be willing and able to comply with the protocol requirements, including the specified Prohibitions and Restrictions.
9. Participant must be willing to provide verifiable identification.
10. Participant must have a means to be contacted. In addition, the participant must be; (1) intending to remain in the study area for the duration of the study (two years) for Ugandan nationals (2) intending to remain in Uganda for international staff for at least 65 days and able to be followed for the duration of the study (two years).

9. Participant must pass the test of understanding/comprehension (TOU) Additional Inclusion Criteria for HIV-infected Participants

All of the inclusion criteria above must be met by adults who are HIV-infected with the following additions/clarifications:

1. Participant must have a documented HIV-infection for at least 6 months prior to screening.
2. Participant must be on a stable regimen of Highly Active Antiretroviral Therapy (HAART), taking into account the following criteria:

   1. HAART is defined as potent anti-HIV treatment including a combination of ≥3 antiretroviral agents (ARVs; low-dose ritonavir does not count as an ARV) whose purpose is to reduce viral load to undetectable levels. Mono- or bitherapy will not be allowed.
   2. HAART is considered stable if participants did not change their ARVs within the last 4 consecutive weeks prior to start of screening. Changes in formulations are allowed.
   3. Participant's medical history (and/or medical records) should demonstrate evidence of immunological stability (CD4+ Tcell count of at least 350 cells/ml within the last 6 months) and HIV virologic control
   4. Participant must be willing to continue their HAART throughout the study as directed by their local physician.
3. Participant must be in an otherwise reasonably good medical condition (absence of acquired immunodeficiency syndrome (AIDS)-defining illnesses or clinically significant disease), diagnosed on the basis of physical examination, medical history and the investigator's clinical judgment.

Exclusion Criteria Any potential participant who meets any of the following criteria will be excluded from participating in the study.

1. Has received any candidate Ebola vaccine in the past.
2. Previously diagnosed with Ebola virus disease (self-report or laboratory confirmed)
3. Has received any experimental candidate Ad26- or MVA-based vaccine in the past. Note: Receipt of any approved vaccinia/smallpox vaccine or Ad-based candidate vaccine other than Ad26 at any time prior to study entry is allowed.
4. Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccines [eg, polysorbate 80, ethylenediaminetetraacetic acid (EDTA) or L-histidine for Ad26.ZEBOV vaccine; tris (hydroxymethyl)-amino methane (THAM) for MVA-BN-Filo vaccine]), including known allergy to egg, egg products and aminoglycosides.
5. Participants with acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or body temperature ≥38.0ºC on Day 1 will be excluded from enrollment at that time, but may be rescheduled for enrollment at a later date.
6. A woman who is pregnant, breast-feeding or planning to become pregnant while enrolled in the study or within at least 3 months after the first vaccination, up to 1 month after the second vaccination (whichever takes longer).
7. Presence of significant conditions (eg, history of seizure disorders, active malignancy, psychiatric or metabolic disturbances) or clinically significant findings during screening of medical history, physical examination, vital signs or laboratory testing for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg, compromise the safety or well-being) or that could prevent, limit, or confound the protocol-specified assessments.
8. Received an investigational drug or investigational vaccine or used an invasive investigational medical device within 3 months prior to screening, or current or planned participation in another clinical study during the study.

   Note: Participation in an observational clinical study is allowed.
9. Receipt of blood products or immunoglobulin within 3 months prior to screening and during participation in the study.
10. Current or past abuse of alcohol, recreational or narcotic drugs, which in the investigator's opinion would compromise the participant's safety and/or compliance with the study procedures.
11. History of chronic urticaria (recurrent hives).
12. Participant cannot communicate reliably with the investigator.
13. Participant who, in the opinion of the investigator, is unlikely to adhere to the requirements of the study.
14. Employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator.
15. History of having received lengthy systemic immunosuppressant therapies (consecutive duration of at least 2 weeks) that would substantially interfere with the mode of action of the Ebola vaccine in the previous 6 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
The total IgG against EBOV-GP at day 77 post-vaccination with Ad26.ZEBOV (dose 1) at day 0 and MVA-BN®-Filo (dose 2) at day 56. | 21-days post second vaccination
  Humoral immune responses as measured by enzyme-linked immunosorbent assay (ELISA) to the Ebola glycoprotein after intramuscular administration of Ad26.ZEBOV/ MVA-BN®-Filo vaccine in all participants on Day 0 and Day 77.
Frequency, incidence and nature of Serious Adverse Events, 6 months following the second vaccination | 6 months following second vaccination
  The occurrence, incidence and nature of Serious Adverse Events between the time of vaccination with Ad26.ZEBOV and during the ¬ 6 months following vaccination with MVA-BN®-Filo. If a participant does not receive MVA-BN®-Filo for any given reason, the outcome will be the occurrence, incidence and nature of SAE during the 6 months following vaccination with Ad26.ZEBOV

SECONDARY OUTCOMES:
The total IgG against EBOV-GP at 365-days post-vaccination with Ad26.ZEBOV/MVA-BN®-Filo | 365-days post-vaccination with Ad26.ZEBOV/MVA-BN®-Filo
  Humoral immune responses as measured by enzyme-linked immunosorbent assay (ELISA) against Ebola glycoprotein after intramuscular administration of Ad26.ZEBOV/ MVA-BN®-Filo vaccine in a subset of participants on Day 365.
The total IgG against EBOV-GP at day 56 | Day 56 post vaccination with Ad26.ZEBOV
  Humoral immune responses as measured by enzyme-linked immunosorbent assay (ELISA) against Ebola glycoprotein after intramuscular administration of Ad26.ZEBOV vaccine in a subset of participants on Day 56
The existing knowledge about Ebola disease and transmission, and the perception and attitudes about the vaccine and protection in a subset of participants. | At baseline (Day 0) and after the second Vaccination
  To describe the knowledge about Ebola virus disease and transmission, and the perception and attitudes about the vaccine and protection in a subset of participants in the Ad26.ZEBOV/MVA-BN®-Filo vaccine study.

OTHER OUTCOMES:
The sero-prevalence of Ebola Zaire, Bundibugyo, Sudan and Marburg specific antibodies | Baseline (Day 0)
  The sero-prevalence of Ebola Zaire, Bundibugyo, Sudan and Marburg specific antibodies as determined by IgG Elisa in all participants
The number of staff trained in Peripheral Blood Mononuclear Cell (PBMC) processing and cryopreservation at Epicentre, Mbarara | During the study
  The Epicentre Mbarara laboratory staff are to be trained in Peripheral Blood Mononuclear Cell (PBMC) isolation and cryopreservation.
Induced plasma cytokines/chemokines as measured by Luminex. | Day 0, 1 and 3 following the first vaccine
  Plasma cytokines/chemokines including IP-10, MIP-1α, MIP-1β, MCP-1, IFN-α2, IFN-gama, IL-1β, IL-1RA, IL-2, IL-4, IL-6, IL-12, IL-18, TNF-α, Lymphotoxin, will be measured using commercial multiplex kits, following manufacturer's instructions. A Luminex 200 analyser with Bio-Plex Manager software will be used to read the plates and determine analyte concentrations.
Induced plasma cytokines/chemokines as measured by Luminex | Day 56, 57 and 59 following the second vaccine
  Plasma cytokines/chemokines including IP-10, MIP-1α, MIP-1β, MCP-1, IFN-α2, IFN-gama, IL-1β, IL-1RA, IL-2, IL-4, IL-6, IL-12, IL-18, TNF-α, Lymphotoxin, will be measured using commercial multiplex kits, following manufacturer's instructions. A Luminex 200 analyser with Bio-Plex Manager software will be used to read the plates and determine analyte concentrations.
To explore T cell mediated responses to the Ad26.ZEBOV/ MVA-BN®-Filo vaccine at baseline and day 77 in a subset of 100 participants | Day 0 and Day 77 post vaccination with MVA-BN-Filo
  The T cell mediated responses to the Ad26.ZEBOV/ MVA-BN®-Filo vaccine at baseline and day 77 in a subset of participants will be measured by the percentage of memory CD4 and CD8 T cells responding to Ebola GP and NP peptides by production of IFN-gamma and/or IL-2 and/or TNF-α in a flow cytometry ICS assay.
The cumulative incidence of laboratory-confirmed Ebola virus disease cases among eligible persons from first vaccination until study end | Througout the trial and in case of an outbreak
  Laboratory confirmed EVD cases defined as: Any probable or suspected case from which a blood sample taken is laboratory confirmed as positive for EVD; or, Any deceased individual with probable EVD, from which a post-mortem sample taken within 48 hours after death is laboratory confirmed as positive for EVD. Laboratory confirmation is by validated real-time reverse transcriptase (RT) PCR-based assay for Ebola viral nucleic acid.

CONTACTS AND LOCATIONS:
Locations (1):
- MRC/UVRI & LSHTM Uganda Research Unit, Entebbe, Uganda

IPD SHARING:
Plan to Share IPD: No